CLINICAL TRIAL: NCT06461793
Title: Safety of Dose Escalation in Definitive Hypofractionated Radiation Therapy and Hormone Therapy With SpaceOAR TM for Patients With High - Risk Localized Prostate Cancer (DESAR-H)
Acronym: DESAR-H
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Park, Won Park, M.D., Ph.D., Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2023-06-140
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: High Risk Prostate Carcinoma

STUDY DESIGN:
Intervention Model Description: - A single institution with a single group, a phase II study, we plan to evaluate grade 1 or higher rectal bleeding within 3 years in high-risk prostate cancer patients who received biodegradable substance injection followed by curative radiotherapy in combination with hormone therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate cancer patient, candidate of definitive radiation treatment (Experimental): A single institution with a single group, a phase II study, we plan to evaluate grade 1 or higher rectal bleeding within 3 years in high-risk prostate cancer patients who received biodegradable substance injection followed by curative radiotherapy in combination with hormone therapy.
  Interventions: Radiation: Dose increase after injection of biodegradable material A safety study of high-risk prostate cancer patients

INTERVENTIONS:
Radiation: Dose increase after injection of biodegradable material A safety study of high-risk prostate cancer patients — this researcher performed biodegradable material injection during radical radiotherapy in combination with hormone therapy in high - risk prostate cancer patients. after subdivision radical received radiation therapy We plan to conduct a phase II clinical study to evaluate the safety of prostate cancer patients.

SUMMARY:
Dose increase after injection of biodegradable material A safety study of high-risk prostate cancer patients who underwent low-fractionation curative radiation therapy and hormone therapy

DETAILED DESCRIPTION:
In prostate cancer, radiation therapy for curative purposes can be used regardless of the stage if there is no distant metastasis, and radiation therapy and hormone therapy may be combined in patients with moderate or high risk factors for recurrence. Randomized prospective studies to investigate the therapeutic effect of increasing dose escalation to 70 Gy or more showed significant reductions in biochemical failure. When the dose is increased, the risk of side effects (digestive system, urinary system) in surrounding normal tissues increases, and intensity modulated radiation therapy (IMRT) or image-guided radiation therapy (IGRT) Application could reduce the probability of side effects. Prostate cancer is a carcinoma characterized by slow growth, and the estimated α/β ratio is 1.5, which is smaller than surrounding normal tissues such as the bladder (4.0) and the rectum (3.9). Therefore, efforts to obtain therapeutic gain through hypofractionated radiation therapy have been attempted using three-dimensional conformal radiotherapy (3D-CRT) and IMRT. In particular, in the CHHIP trial11 announced in 2016, normal division Radiation therapy (74 Gy, 37 splits ) and as a result of comparing low-fractionation radiation therapy (60 Gy, 20 fractions ), there was no significant difference in the 5 -year biochemical or clinical recurrence -free survival rate of low-fractionation radiation therapy, it was also reported that there was no difference in rectal and bladder side effects. However, rectal and bladder side effects of grade 2 or higher were 11.9% and 11.7 % during one-time 3 Gy low-fractionated radiotherapy, respectively. The low-fractionated radiotherapy dose is 81 Gy, which is the recommended normal fractionated radiotherapy dose when using IMRT. It can be said that there is a high possibility of showing inferior treatment results in long-term follow-up results because the biological effective dose is lower than that of 'ideal '. ( Table 1)

* Table 1. Biological Equivalent Dose by Radiation Therapy Policy (2-Gy fraction) comparison
* Protocol: EQD1 (Gy)(α/β=1.5)
* Low-fraction radiation therapy (70 Gy, 28 sessions): 80.0 Gy
* Conventional fractionation radiation therapy (74 Gy, 37 times): 74 Gy
* CHHIP trial (60 Gy, 20 times): 77.14 Gy
* study design dose(64 Gy, 20 times): 85.94 Gy *EQD2, equivalent dose in 2-Gy fractions

Recently , a method was devised to increase the distance between prostate and rectum by injecting hydrogel between prostate and rectum to minimize rectal dose even when performing high-dose radiotherapy to prostate. In particular , a biodegradable material ( SpaceOAR (hydrogel)) that is absorbed into the body after a certain period of time has been developed, and radical radiation therapy is performed. It is currently being used in prostate cancer patients. It is judged possible to try to increase the radiation dose because the side effects can be reduced by reducing the rectal dose during radical radiation treatment through biodegradable material injection. So far, studies evaluating the side effects of treatment according to increased radiation dose after injection of biodegradable materials are very limited. Therefore, the investigator performs biodegradable material injection before radical radiotherapy in combination with hormone therapy in high - risk prostate cancer patients. The investigator plans to conduct a phase II clinical study to evaluate the safety of high - risk prostate cancer patients who has received subdivision radical radiation therapy with hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed prostate adenocarcinoma within 6 months of study enrollment
2. Patients with prostate cancer at high risk or above (c T3a-T4 or grade group 4-5 or PSA > 20 n g/mL) )
3. Patients who have undergone or are scheduled to undergo hormone therapy for high-risk prostate cancer
4. Adults over 20 years of age
5. Whole body performance ECOG 0-1
6. SpaceOAR Patients who consented to the procedure and study

Exclusion Criteria:

1. prostate removal surgery, Patients with a history of lower pelvic surgery including rectal cancer surgery
2. primary cancer Patients with posterior extracapsular extension
3. Medically biodegradable substances such as bleeding predisposition Patients for whom infusion is not appropriate
4. Patients with a history of previous pelvic radiation therapy
5. Patients with lymph node metastasis or distant metastasis

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Histopathologically confirmed prostate adenocarcinoma within 6 months of study enrollment
Enrollment: 33 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
NIH-NCI Common Terminology Criteria for Adverse Events (CTCAE) V 5.0 Frequency of rectal bleeding of grade 1 or higher within 3 years | 3 years after radiation therapy of each participant
  Adverse Event within three years after the radiation therapy

SECONDARY OUTCOMES:
Radiation therapy-related side effects other than rectal bleeding | up to 2 years afte radiation therapy on each participant
  Sigmoi doscopy is performed once a year for up to 2 years after the end of radiation therapy,
Side effects related to biodegradable material injection | each participant finished with radiation therapy and see after 3-6 months for acute adverse events, 1-5 years for chronic adverse events
biochemical recurrence-free survival | 5 years after radiation therapy of each participant
  Biochemical recurrence is defined as PSA nadir + 2.0ng/ml according to the Phoenix definition, or when hormone therapy is discontinued, when hormone therapy is newly started, or when hormone therapy is in progress, when the treatment is changed.
progression-free survival | up to 5 years after radiation therapy of each participant
  check on each participant by CT scan, MRI, Bone scan for any progressive disease
overall survival | up to 5 years after radiation therapy of each participant
  overall survival of participants till the end of the study(death)
quality of life on high-risk prostate cancer patients by using EPIC questionnaire | up to 5 years after radiation therapy of each participant
  EPIC (Extended Prostate Cancer Index Composite), Korean version

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: SpaceOAR™ Hydrogel is Associated with Lower Rectal Toxicity and Higher Bowel Quality of Life in Late Follow-up: Systematic Review & Meta-Analysis — https://www.bostonscientific.com/content/dam/bostonscientific/spaceoar/vue/infographic-spaceoar-hydrogel-meta-analysis.pdf